CLINICAL TRIAL: NCT00417469
Title: A Single-Blind, Randomized, Single-Center Evaluation of Procedural and Post Procedural Pain Experienced With Injections of NADG With Lidocaine Injectable Gel as Compared to Captique® Injectable Gel in Subjects Undergoing Cutaneous Correction of Nasolabial Folds
Brief Title: A Study to Compare Subject Comfort During and After Injections With the Study Products and the Safety of the Non-FDA Approved Product for the Correction of Nasolabial Folds (NLFs)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: NADGL00106
Record Dates: First submitted 2006-12-28; First posted 2007-01-01 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Facial Wrinkles

STUDY DESIGN:
Who Masked: Participant

INTERVENTIONS:
Device: NADGL

SUMMARY:
The purpose of this research study is to compare subject comfort during and after injection with NADGL and Captique® Injectable Gel, in the nasolabial folds. Captique® is an FDA-approved product without lidocaine and is manufactured by Genzyme Biosurgery (Ridgefield, NJ). NADGL is a new product (not FDA approved) with lidocaine and is also manufactured by Genzyme Biosurgery. We do not know which of these treatments results in less pain during and after injection. The safety of NADGL is also being studied.

DETAILED DESCRIPTION:
45 subjects are planned; a portion of these subjects will have skin of color

ELIGIBILITY:
Inclusion Criteria:

* bilateral nasolabial folds with severity score of 3 or 4 on the 6 point scale.

Exclusion Criteria:

* pregnant/lactating women
* subjects who have an allergy to lidocaine or other amide-type anesthetics

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 45
Dates: Start 2007-01; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the pain experienced during and after the injection procedure for NADGL as compared to Captique® Injectable Gel in subjects undergoing cutaneous correction of nasolabial folds (NLFs).

SECONDARY OUTCOMES:
To evaluate the safety of NADGL.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (1):
- Birmingham, Alabama, United States